CLINICAL TRIAL: NCT02554136
Title: An Open-labeled, Randomized Crossover Study to Evaluate the Pharmacokinetic Interaction and Safety After Single Oral Administration of HGP0918 and HGP0816 in Healthy Adult Subjects
Brief Title: Evaluating a Pharmacokinetic Drug Interaction Between HGP0918 and HGP0816
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ROMA-105
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental): HGP0918 -> HGP0816 -> HGP0918 + HGP0816
  Interventions: Drug: HGP0918; Drug: HGP0816; Drug: HGP0918 + HGP0816
- Sequence 2 (Experimental): HGP0816 -> HGP0918 + HGP0816 -> HGP0918
  Interventions: Drug: HGP0918; Drug: HGP0816; Drug: HGP0918 + HGP0816
- Sequence 3 (Experimental): HGP0918 + HGP0816 -> HGP0918 -> HGP0816
  Interventions: Drug: HGP0918; Drug: HGP0816; Drug: HGP0918 + HGP0816
- Sequence 4 (Experimental): HGP0918 -> HGP0918 + HGP0816 -> HGP0816
  Interventions: Drug: HGP0918; Drug: HGP0816; Drug: HGP0918 + HGP0816
- Sequence 5 (Experimental): HGP0816 -> HGP0918 -> HGP0918 + HGP0816
  Interventions: Drug: HGP0918; Drug: HGP0816; Drug: HGP0918 + HGP0816
- Sequence 6 (Experimental): HGP0918 + HGP0816 -> HGP0816 -> HGP0918
  Interventions: Drug: HGP0918; Drug: HGP0816; Drug: HGP0918 + HGP0816

INTERVENTIONS:
Drug: HGP0918
Drug: HGP0816
Drug: HGP0918 + HGP0816

SUMMARY:
The investigators investigate the potential pharmacokinetic drug-drug interaction between HGP0918 and HGP0816 in healthy adult subjects who receive HGP0918 alone, HGP0816 alone, and both together in a 3 period repeatedly

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing
* Healthy male volunteers, aged 19 to 55 years.
* The result of Body Mass Index(BMI) is not less than 18.5 kg/m2 , no more than 27.0 kg/m2

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
* Someone has a declined liver function and Liver enzyme (AST, ALT or total bilirubin) level exceeds more than one and a half times normal upper range
* Somenone has a declined kidney function and his eGFR < 60mL/min/1.73m2

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
baseline-corrected Cmax of HGP0918 | -20, -16, -12, 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72hr (Total 16)
baseline-corrected AUCt of HGP0918 | -20, -16, -12, 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72hr (Total 16)
Cmax of HGP0816 | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)
AUCt of HGP0816 | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)

SECONDARY OUTCOMES:
Cmax of HGP0918 | -20, -16, -12, 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72hr (Total 16)
AUCt of HGP0918 | -20, -16, -12, 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72hr (Total 16)
Tmax of HGP0918 | -20, -16, -12, 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72hr (Total 16)
t1/2β of HGP0918 | -20, -16, -12, 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72hr (Total 16)
AUC∞ of HGP0816 | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)
Tmax of HGP0816 | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)
t1/2β of HGP0816 | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)
CL/F of HGP0816 | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)
Vdz/F of HGP0816 | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)

CONTACTS AND LOCATIONS:
Locations (1):
- Inje Busan Paik hospital, Busan, South Korea